CLINICAL TRIAL: NCT04537689
Title: Outcomes With Treatment and Withdraw of Ixekizumab in Patients With Plaque Psoriasis Compared to Standard Care --- a Pragmatic Observational Study
Brief Title: Outcomes With Treatment and Withdraw of Ixekizumab in Patients With Plaque Psoriasis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Translational Immunology Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PsO_IXE
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — ixekizumab; Methotrexate; Cyclosporine; Acitretin

STUDY DESIGN:
Intervention Model Description: To evaluate the real-life effectiveness of ixekizumab as first-line systemic treatment in participants with moderate to severe PsO, the investigators would recruit a pragmatic control arm.
  ⦁ Intervention arm: Eligible participants will be offered ixekizumab as first-line systemic treatment for PsO. Standard dose of subcutaneous ixekizumab for moderate to severe PsO will be given at 160 mg at week 0, followed by ixekizumab 80mg at weeks 2, 4, 6, 8, 10 and 12, then 4 weekly thereafter, for a total duration of 6 months.
  Ixekizumab will be withdrawn after 6 months. For some participants, there may be relapse of PsO. Relapses will be managed as per standard care.
  ⦁ Pragmatic control arm
  Eligible participants will be recruited to pragmatic control arm in these circumstances:
  * Patient disagree to ixekizumab for personal reasons.
  * The quota for ixekizumab is exhausted.
  * The management of PsO in this pragmatic control arm will be the same as that in the standard care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ixekizumab (Experimental): Participants will be offered ixekizumab as first-line systemic treatment for moderate to severe PsO. The indication for ixekizumab will be equivalent to current registered indications. Standard dose of subcutaneous ixekizumab for moderate to severe PsO will be given at 160 mg at week 0, followed by ixekizumab 80mg at weeks 2, 4, 6, 8, 10 and 12, then 4 weekly thereafter, for a total duration of 6 months.
  Ixekizumab will be withdrawn after 6 months. For some participants, there may be relapse of PsO.
  Relapses will be managed as per standard care.
  Interventions: Biological: Ixekizumab
- Standard Care (Active Comparator): The management of PsO in the control arm will be the same as that in the standard care.
  The standard care for moderate to severe PsO in Singapore is to start either phototherapy, methotrexate, acitretin or cyclosporin A.
  Interventions: Drug: Methotrexate; Drug: Cyclosporin A; Drug: Acitretin

INTERVENTIONS:
Biological: Ixekizumab — Ixekizumab for 6 months, given 160mg at weeks 0, followed by 80mg at 2, 4, 6, 8, 10 and 12, then 4 weekly till 6 months. Given subcutaneously.
  Arms: Ixekizumab
Drug: Methotrexate — Oral tablet up to 15mg per week
  Arms: Standard Care
Drug: Cyclosporin A — Oral capsule up to 200mg per day
  Arms: Standard Care
Drug: Acitretin — Oral capsule up to 25mg per day
  Arms: Standard Care

SUMMARY:
Psoriasis (PsO) is a systemic immune disease that affect 2-4% of the population worldwide. PsO causes tremendous burden in terms of quality of life, psychological impact, disability and work productivity of affected individuals. PsO is associated with an increased risk of cardiovascular morbidities and mortality in the long term. Up to 30% of PsO patients develop psoriatic arthritis (PsA) over time causing joint deformities and further disabilities. Majority of patients with PsA developed PsO first, and arthritis develop 5-10 years afterwards. PsA and PsO are increasingly recognized as two entities under the umbrella of psoriatic diseases.

Advances in biological treatments have greatly improved the prognosis of patients with PsO. Remarkable efficacies have been demonstrated for patients with moderate to severe PsO in randomized controlled trials (RCTs). However, the high cost of biological treatment is one of the major barriers to prescription of biological treatment and many patients may have limited access to these treatments.

The best strategy of treatment for PsO that takes into account efficacy and cost effectiveness is unknown. For instance, whether some PsO patients can stop biological treatment and be retreated with non-biologic medications upon relapse, which may enhance cost effectiveness of treatment. Preliminary studies have shown that some PsO patients were able to maintain good control of disease without medications after biologics withdrawal. The patho-immunological mechanisms behind long term remission after drug withdrawal is poorly understood. Better understanding on patho-immunological mechanisms on maintenance of remission and relapses will advance the development of biomarkers that eventually guide development of best treatment strategies for PsO.

Ixekizumab is a humanized immunoglobulin G4 (IgG4 kappa) monoclonal antibody targeting interleukin (IL)-17A. It is highly efficacious in the treatment of plague PsO with and favorable safety profile as shown in randomized controlled trials, and is an approved treatment for moderate-to-severe PsO by the U.S. Food and Drug Administration and Health Sciences Authority. With the proven efficacies, ixekizumab could be a choice of first-line treatment for patients with moderate to severe PsO. The 2013 American Academy of Dermatology position statement have stated that the old paradigm of stepwise-therapy starting first with phototherapy and oral systemic therapies before biologic treatment is not required for patients with moderate to severe PsO. In the recent 2017 update of the European S3 guidelines also recommend the use of IL-17 inhibitors as either a first- or second-line agent. In a RCT that evaluated relapses after withdrawal of ixekizumab among patients who achieved a clearance of PsO, loss of PsO clearance were seen after a median of 20 weeks. Response can be successfully recaptured in over 80% of patients with retreatment with ixekizumab, suggesting that the treatment regimen could be interrupted in some patients. However, real-life data on biologic treatment or withdrawal for moderate to severe PsO is scatty.

DETAILED DESCRIPTION:
First, the investigators hypothesize that a proportion of patients with moderate to severe PsO may sustain reasonable good outcomes when a short course of ixekizumab is withdrawn.

Second, the investigators hypothesize that the investigators can identify the perturbations in the architecture of the immunome which are pathogenic, and to discriminate such perturbations based on treatment and clinical responses, thus distilling theragnostic signatures.

Therefore, the objectives of the study are as follow:

Specific aim 1: To describe the clinical course, sustained good outcomes, relapse rate, time to relapse and quality of life in PsO patients who stopped a 6-month short course treatment of ixekizumab, till the end of 2-years.

Specific aim 2: To identify the genomic and immunomic signatures in skin biopsies and blood in PsO patients who has good outcomes (PASI 75) at 6 months, comparing treatment vs pragmatic control.

Specific aim 3: To identify the genomic and immunomic signatures in skin biopsies and blood in PsO patients who sustained good outcomes at 1 year after stopping ixekizumab, compared to those relapsed.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>21-year-old).
* Diagnosed by dermatologist as plague-type PsO.
* Having moderate to severe plague-type PsO as defined by the following:
* Psoriasis Area and Severity Index (PASI) ≥12/72,
* And, investigator Global Assessment Score (IGA) ≥3,
* And, PsO involving body surface area involvement (BSA) ≥10%
* And Candidate for phototherapy and/or systemic therapy
* Topical corticosteroid up to moderate potencies are allowed
* Able to provide informed consent.

Exclusion Criteria:

* Forms of PsO other than plaque-type.
* Evidence of skin conditions at the time of the screening visit (e.g. eczema) that would interfere with evaluation of the effect of the investigational product on PsO.
* Evidence of active tuberculosis or other active infections (like Hepatitis C/B), malignancy; active or known use of other immunosuppressive drugs (eg. AIDS, rheumatoid arthritis, organ rejection etc) at the screening visit.
* Previous exposure to any systemic immunosuppressants (eg. methotrexate) or phototherapy
* History or current signs of a severe, progressive, or uncontrolled renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances.
* Having current or history of malignancy, except non-melanoma skin cancer, within the previous 5 years that have been adequately treated.
* History of inflammatory bowel disease.
* Pregnancy or lactating mothers.
* As treatment regimen is different, participants with evidence of PsA will be excluded

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of ixekizumab treated PsO participants free of relapse after ixekizumab withdrawal | 12 months from ixekizumab withdrawal or 18 months from baseline.
  The investigators will describe the proportion of ixekizumab treated PsO participants free of relapse at 12 months after ixekizumab withdrawal.

SECONDARY OUTCOMES:
Proportion of ixekizumab treated PsO participants free of relapse after ixekizumab withdrawal | 15, 18, and 24 months from ixekizumab withdrawal or 21, 24, and 30 months from baseline.
  The investigators will describe the proportion of ixekizumab treated PsO participants free of relapse at 15, 18, and 24 months after ixekizumab withdrawal.
Proportion of participants achieving PASI 50 | 3 months and 6 months
  Psoriasis is assessed by using the Psoriasis Area Severity Index (PASI) that measures the severity (intensity of redness, thickness and scaling is assessed as none (0), mild (1), moderate (2), severe (3) or very severe (4)) and percentage of affected area in four regions of the body (head and neck, upper limbs, trunk, lower limbs, expressed as nil (0), 1-9% (1), 10-29% (2), 30-49% (3), 50-69% (4), 70-89% (5) or 90-100% (6)). The score ranges from 0 (no psoriasis) to 72 (severe psoriasis). Percentage of improvement of PASI at 3 month and 6 month time points will be calculated from baseline. PASI 50 indicates a 50% improvement of PASI scores.
Proportion of participants achieving PASI 75 | 3 months and 6 months
  Psoriasis is assessed by using the Psoriasis Area Severity Index (PASI) that measures the severity (intensity of redness, thickness and scaling is assessed as none (0), mild (1), moderate (2), severe (3) or very severe (4)) and percentage of affected area in four regions of the body (head and neck, upper limbs, trunk, lower limbs, expressed as nil (0), 1-9% (1), 10-29% (2), 30-49% (3), 50-69% (4), 70-89% (5) or 90-100% (6)). The score ranges from 0 (no psoriasis) to 72 (severe psoriasis). Percentage of improvement of PASI at 3 month and 6 month time points will be calculated from baseline. PASI 75 indicates a 75% improvement of PASI scores.
Proportion of participants achieving PASI 90 | 3 months and 6 months
  Psoriasis is assessed by using the Psoriasis Area Severity Index (PASI) that measures the severity (intensity of redness, thickness and scaling is assessed as none (0), mild (1), moderate (2), severe (3) or very severe (4)) and percentage of affected area in four regions of the body (head and neck, upper limbs, trunk, lower limbs, expressed as nil (0), 1-9% (1), 10-29% (2), 30-49% (3), 50-69% (4), 70-89% (5) or 90-100% (6)). The score ranges from 0 (no psoriasis) to 72 (severe psoriasis). Percentage of improvement of PASI at 3 month and 6 month time points will be calculated from baseline. PASI 90 indicates a 90% improvement of PASI scores.
Proportion of participants achieving clearance | 3 months and 6 months
  Psoriasis is assessed by using the Psoriasis Area Severity Index (PASI) that measures the severity (intensity of redness, thickness and scaling is assessed as none (0), mild (1), moderate (2), severe (3) or very severe (4)) and percentage of affected area in four regions of the body (head and neck, upper limbs, trunk, lower limbs, expressed as nil (0), 1-9% (1), 10-29% (2), 30-49% (3), 50-69% (4), 70-89% (5) or 90-100% (6)). The score ranges from 0 (no psoriasis) to 72 (severe psoriasis). Percentage of improvement of PASI at 3 month and 6 month time points will be calculated from baseline. Clearance indicates a 100% improvement of PASI scores.
Quality of life 1 (EuroQoL-5D-5L) | 3, 6, 9, 12, 15, 18, 24 and 30 months
  In all participants (both ixekizumab treated and standard care) the investigators will describe the following:
  Every 3-6 monthly till end of 30 months, investigators will evaluate the change scores of Quality of Life (EQ5D-5L). It consists of the EQ-5D-5L descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions. Each dimension is measured on a scale of 1-5, with '1' indicating no problem, '2' indicating slight problems, '3' indicating moderate problems, '4' indicating severe problems, and '5' indicating unable to/extreme problems. The highest and the lowest scores for both EQ-5D-5L indices were 1.00 (best imaginable health) and -0.769 respectively; where negative values are valued as worse than dead.
  EQ VAS records the patient's self-rated health on a vertical visual analogue scale from 0-100 with '0' indicating worst health one can imagine and '100' indicating best health one can imagine.
Quality of life 2 (Dermatology Life Quality Index - DLQI) | 3, 6, 9, 12, 15, 18, 24 and 30 months
  In all participants (both ixekizumab treated and standard care) the investigators will describe the following:
  - Questionnaires on health status and quality of life every 3-6 monthly till end of 30 months.
  The investigators will evaluate the change scores of Dermatology Life Quality Index (DLQI) at various time points from baseline. DLQI is measured on a scale of 0-3 or not relevant, with '0' indicating not relevant or not at all, '1' indicating a little, '2' indicating a lot, '3' indicating very much. The final score ranges from 0 (minimal effect on quality of life) to 30 (maximum effect on quality of life).
Quality of life 3 (Hospital Anxiety and Depression Scale - HADS) | 3, 6, 9, 12, 15, 18, 24 and 30 months
  n all participants (both ixekizumab treated and standard care) the investigators will describe the following:
  - Questionnaires on health status and quality of life every 3-6 monthly till end of 30 months.
  The investigators will evaluate the change scores of Hospital Anxiety and Depression Scale (HADS) at various time points from baseline. HADS is a 14 item scale with 7 of the items related to anxiety and the other 7 related to depression. Each item on the questionnaire is scored from 0-3, resulting in anxiety and depression scores each of 0 (no anxiety/depression) to 21 (severe anxiety/depression).
Patient Global Assessment | 3, 6, 9, 12, 15, 18, 24 and 30 months
  In all participants (both ixekizumab treated and standard care) the investigators will describe the following:
  - Questionnaires on health status and quality of life every 3-6 monthly till end of 30 months.
  The investigators will evaluate the change scores of Patient Global Assessment (0-10) at various time points from baseline, with higher scores meaning worse outcome.
Patient Acceptable Symptom State (PASS) | 3, 6, 9, 12, 15, 18, 24 and 30 months
  In all participants (both ixekizumab treated and standard care) the investigators will describe the following:
  - Questionnaires on health status and quality of life every 3-6 monthly till end of 30 months.
  The investigators will evaluate the proportion of patient defined acceptable state (acceptable/unacceptable) and whether the symptoms are worse than usual (yes/no) at various time points from baseline.
Proportion of participants in ixekizumab treatment arm maintaining PASI 50 after ixekizumab withdrawal | 9, 12, 18, 24 and 30 months from baseline
  For participants in the ixekizumab treatment arm, the investigators describe the following in additional:
  - The proportion of participants maintaining PASI 50 at 3, 6, 12, 18 and 24 months after stopping ixekizumab treatment
Proportion of participants in ixekizumab treatment arm maintaining PASI 75 after ixekizumab withdrawal | 9, 12, 18, 24 and 30 months from baseline
  For participants in the ixekizumab treatment arm, the investigators describe the following in additional:
  - The proportion of participants maintaining PASI 75 at 3, 6, 12, 18 and 24 months after stopping ixekizumab treatment
Proportion of participants in ixekizumab treatment arm maintaining PASI 90 after ixekizumab withdrawal | 9, 12, 18, 24 and 30 months from baseline
  For participants in the ixekizumab treatment arm, the investigators describe the following in additional:
  - The proportion of participants maintaining PASI 90 at 3, 6, 12, 18 and 24 months after stopping ixekizumab treatment
Proportion of participants in ixekizumab treatment arm maintaining clearance after ixekizumab withdrawal | 9, 12, 18, 24 and 30 months from baseline
  For participants in the ixekizumab treatment arm, the investigators describe the following in additional:
  - The proportion of participants maintaining PASI clearance at 3, 6, 12, 18 and 24 months after stopping ixekizumab treatment
Proportion of participants in ixekizumab treatment arm flaring after ixekizumab withdrawal | 9, 12, 18, 24 and 30 months from baseline
  For participants in the ixekizumab treatment arm, the investigators describe the following in additional:
  - The proportion of participants who flare (defined as losing the PASI50 response) at 3, 6, 12, 18 and 24 months after stopping ixekizumab treatment
Histological changes in the skin biopsies of participants in ixekizumab treatment arm who relapsed after ixekizumab withdrawal (or at 18 months if no relapse) | Baseline, 6 months, at relapse (or 18 months if no relapse)
  For participants in the ixekizumab treatment arm, the investigators will evaluate the following outcomes at relapse (or at 12 months after stopping ixekizumab if no relapse):
  - Histological sections of morphologically psoriasis (lesional) and morphologically no psoriasis (nonlesional) skin biopsies. Skin biopsies at relapse will be scored for the degree of histological improvement compared to that participant's disease at 6 months on a five point scale; -1 (worse) to +3 (excellent).
Skin genomic profiles in the skin biopsies of participants in ixekizumab treatment arm who relapsed after ixekizumab withdrawal (or at 18 months if no relapse) | Baseline, 6 months, at relapse (or 18 months if no relapse)
  For participants in the ixekizumab treatment arm, the investigators will evaluate the following outcomes at relapse (or at 12 months after stopping ixekizumab if no relapse):
  - Whole RNA genome transcriptome of the skin biopsies will be studied. The change in transcriptomes at relapse compared to 6-month will be evaluated.
Peripheral blood immunome profiles of participants in ixekizumab treatment arm who relapsed after ixekizumab withdrawal (or at 18 months if no relapse) | Baseline, 6 months, at relapse (or 18 months if no relapse)
  For participants in the ixekizumab treatment arm, the investigators will evaluate the following outcomes at relapse (or at 12 months after stopping ixekizumab if no relapse):
  1. The B-cell and T-cell subtypes in the peripheral blood will be evaluated using mass cytometry, and compared to that of baseline and 6 months.
  2. The investigators will evaluate the change in B-cell and T-cell Subtypes at relapse compared to baseline and 6 months.
Histological changes in the skin biopsies | Baseline and 6 months
  In all participants, the investigators will evaluate the skin genomic profiles that differentiate between ixekizumab versus standard care control arms.
  - Histological sections of morphologically psoriasis (lesional) and morphologically no psoriasis (non lesional) skin biopsies at baseline and 6 months will be examined. Skin biopsies at 6 month will be scored for the degree of histological improvement compared to that participant's baseline disease on a five point scale; -1 (worse) to +3 (excellent).
Skin genomic profiles | Baseline and 6 months
  In all participants, the investigators will evaluate the skin genomic profiles that differentiate between ixekizumab versus standard care control arms.
  - Whole RNA genome transcriptome of the skin biopsies will be studied. The change in transcriptomes at 6 months compared to baseline will be evaluated.
Peripheral blood immunome profiles | Baseline and 6 months
  In all participants, the investigators will evaluate the blood immunome profiles that differentiate between ixekizumab versus standard care control arms.
  - The B-cell and T-cell subtypes in the peripheral blood of participants in both ixekizumab and standard care arms will be evaluated using mass cytometry. - The investigators will evaluate the change in B-cell and T-cell subtypes at 6 months from baseline for all participants

CONTACTS AND LOCATIONS:
Overall Officials: Ying Ying Leung, MD, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Outram Park, Singapore

IPD SHARING:
Plan to Share IPD: No